CLINICAL TRIAL: NCT06613607
Title: Effects of Core Strengthening on Pelvic Tilt, Dynamic Balance and Agility in Lower Cross Syndrome: a Quasi-experimental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/29
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: Lower Cross Syndrome

STUDY DESIGN:
Intervention Model Description: Quasi Experimental Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): The group will receive strengthening treatment protocol. Strengthening will be divided into following phases
  1. Warm up phase:
  2. Strengthening phase:
  3. Cool down phase:
  Interventions: Other: Core Strengthening

INTERVENTIONS:
Other: Core Strengthening — Strengthening protocol will comprise of following three phases:
  Warm up phase Following exercise would be performed in warm up; Scissor skier, Criss cross crunches, , Hip circles, Bent over twist.
  Strengthening:
  Abdominal bracing Bracing with heel slides Bracing with leg lifts Bracing with bridging Quadruped alternate arm and leg lifts with bracing Side support with knees flexed Cool down phase: Following exercise would be performed for cood down: Child's pose, Cat cow stretch, Lower back stretch, Obliques stretch

SUMMARY:
This study is a quasi experimental study and the purpose of this study is to determine the effects of core strengthening on pelvic tilt, dynamic balance and agilty in lower cross syndrome.

DETAILED DESCRIPTION:
Participants will be recruited into the study using the criteria of lower crossed syndrome which is assessed using te following tests:

Prone hip extension test Trunk flexion strength test Tightness in erector spinae Modified Thomas test

ELIGIBILITY:
Inclusion Criteria:

* Age 19-35 years
* Both genders
* Positive modified Thomas test
* Positive prone hip extension strength test
* Positive trunk flexion strength test
* Tight erector spinae
* Asia pacific BMI normal (18.5-24.9 Kg/m2)
* Local intermittent lumbar pain
* moderate pain (NPRS 3-7)
* Painless movement and activity
* Pain only produced by sustained loading in relevant position, which is then relieved on moving from that pos

Exclusion criteria:

* Acute flare of LBP
* Centralization and peripheralization of pain
* Signs of stenosis(leg symptoms when walking that are eased upon flexion)
* Pain due to repetitive movements
* Paresthesia/Numbness
* Structual deformity(Kyphosis, spondylosis, spondylolisthesis,scoliosis and joint contractures)
* Curve reversal
* Pregnancy
* Post surgery
* Degenerative and inflammatory spine diseases

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Lumber lordotic angle | 6 weeks
  Lumber lordotic angle will be measured using a mobile applicationOne sensor will be placed at T12- L1 and other sensor will be placed at L5- S1. The sum of these two angles will be calculated.
Dynamic Balance | 6 weeks
  Measured using the star excursion test. It is performed with the subject standing on the middle of the grid on the leg to be tested. The grid consists of 8 lines corresponding to the direction of reach extending out from the center at 45 degrees. The subject will try to reach as far as possible with their feet and the distance from the center will be measured and recorded. This will be repeated 3 times for that direction and performed so for all the directions.
Agility | 6 weeks
  It will be measured using the Illinois agility test, The subject will lie on their front (head to the start line). On the 'Go' command the stopwatch is started, and the subject gets up as quickly as possible and runs forwards 10 meters to run around a cone, then back 10 meters, then runs up and back through a course of four cones. Finally, the athlete runs another 10 meters up and back past the finishing cone, at which the timing is stopped.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan